CLINICAL TRIAL: NCT03350711
Title: A Screening and Recruitment Study in Adults Expressing Interest in the Emory Microbiota Enrichment Program
Acronym: MEP
Status: Suspended | Type: Observational
Why Stopped: The study is temporarily suspended pending additional funding.
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Colleen S. Kraft, Associate Professor, Emory University
Other Study IDs: IRB00098240
Record Dates: First submitted 2017-09-29; First posted 2017-11-22 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Clostridium Difficile Infection
Keywords: Microbiota composition; Microbiota Enrichment Program; Fecal microbiota transplant (FMT)
MeSH Terms: conditions — Clostridium Infections

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Microbiota Enrichment Program (MEP): Patients who are seeking a fecal microbiota transplant (FMT), for any reason, who will be part of a registry of patients to potentially screen for a FMT study.
  Interventions: Other: Microbiota Enrichment Program (MEP)

INTERVENTIONS:
Other: Microbiota Enrichment Program (MEP) — Registry participants will provide demographic and medical information and may take part in general screening procedures to facilitate enrolling into an appropriate FMT study.
  Once determined to be eligible for study entry, study-specific screening procedures may include:
  * Health history and physical examination
  * Urinalysis
  * Urine or serum pregnancy test
  * Blood tests for Hepatitis B, Hepatitis C, HIV, chemistry panel (which includes liver function, kidney function), complete blood count with differential, platelet count, partial thromboplastin time (PTT), international normalized ratio (INR)
  * Electrocardiogram (EKG or ECG)
  * Stool studies
  Participants will be re-screened every 6 months and will remain in follow-up indefinitely or until they are rendered ineligible, participate in a MEP study, or withdraw consent to be included in the database.

SUMMARY:
The goal of this study is to rapidly identify subjects who are eligible for the Microbiota Enrichment Program (MEP) at Emory in Atlanta, Georgia. This general screening protocol will be used to screen potential subjects for the Emory MEP and will be conducted at the Emory Clinic, the Hope Clinic of the Emory Vaccine Center and/or Emory affiliated hospitals. An electronic database will be created to capture demographic and medical information about individuals who are reaching out to obtain fecal microbiota transplant (FMT) and pre-screen these potential study participants for current and upcoming studies within MEP.

DETAILED DESCRIPTION:
The unintended consequence of the development of life-saving antimicrobial therapies has been the havoc that is wreaked on the patient's intestinal microbiota. Clostridium difficile infection (CDI) has been found to be the causative agent of 15%-25% of all cases of antibiotic-associated diarrhea, with increasing severity in those with advanced age and who are hospitalized for other reasons. Despite resolution of symptoms in patients treated with antimicrobials, there remains an ~20% CDI recurrence rate. Furthermore, patients who experience a first recurrence have a 40% risk of an additional recurrence and those with two or more episodes face a 60% risk. As a result, there are substantial numbers of patients who live with chronic and debilitating diarrhea from CDI despite repeated courses of prolonged therapy. C. difficile infection represents an important clinical syndrome and development of new preventive and therapeutic strategies are a key unmet medical need.

Fecal microbiota transplant (FMT), which is defined as the transfer of the feces from one individual (donor) into another individual (recipient), has recently become more standardized and acceptable for the treatment of C. difficile. The first randomized controlled trial (RCT) was published in January of 2013 and compared duodenal infusion FMT after oral vancomycin as compared to oral vancomycin alone and for the treatment of recurrent C. difficile. The trial showed excellent efficacy for FMT, along with restoration of the diversity of the microbiota in the recipients. Even prior to this RCT, case series with over 200 patients had shown excellent efficacy with one FMT, with rates of success almost to 90% when patients received two FMTs.

Emory's Fecal Transplant Program was started in 2012, and since then has performed 280 FMTs in inpatient and outpatient settings. The Emory Microbiota Enrichment Program (MEP) came into existence in 2016 in order to provide a clinical research infrastructure to recruit subjects into clinical research studies related to the microbiome. The goal of this protocol is to create an electronic database capture with a survey to capture demographic and medical information about subjects reaching out to obtain FMT for a variety of reasons and, if needed, pre-screen these subjects for current and upcoming protocols within MEP. A list of potential participants will be generated using the Emory University Data Warehouse to identify subjects with CDI and other conditions that could benefit from the Emory MEP. Advertisements will be placed in the community as a recruitment tool and individuals that contact Emory will be connected to the study recruiter. The recruiters will review the eligibility criteria for inclusion in the MEP database as well as the inclusion and exclusion criteria for all of the enrolling FMT studies currently underway at the Hope Clinic and Emory University Hospitals. If the subject meets the inclusion criteria for one of the Emory FMT studies, they will be invited for a general screening visit or a study specific screening visit for a specific MEP protocol.

The duration of the study varies for each subject and participation is indefinite unless one of the following occurs:

* A subject is rendered ineligible
* The screening is completed, and a subject is referred to a specific MEP study.
* A subject withdraws consent to participate in this study, which may be done verbally or by revocation letter. Additional details will be requested to determine if the participant either no longer wants to perform any MEP related activities (e.g., MEP survey) or revokes the future use of protected health information (PHI) and medical chart review during follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Age of at least 18 years
* Seeking services that are affiliated with the Emory Microbiota Enrichment Program (MEP) for any reason, such as:

  * Clinical services, interventions, or procedures (e.g., FMT), or
  * Research studies
* Able to understand and approve the informed consent and HIPAA authorizations forms verbally on the phone or by signature in-person

Exclusion Criteria:

* Known or suspected terminal disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Recruitment for this study will be done using Emory's data warehouse, subjects with a diagnosis of Clostridium difficile infection (CDI), or subjects that contact Emory with interest in FMT, as well as through referrals from local doctor's offices, and subjects who self-refer to the Emory Microbiota Enrichment Program (MEP)
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2018-09-13 (Actual); Primary Completion 2028-01 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
To determine if the creation of a database will improve enrollment onto other research studies | Ten years
  Successful creation of the database will be defined as capturing demographic and medical information about persons reaching out to obtain FMT in order to screen them for current and upcoming protocols within MEP.

CONTACTS AND LOCATIONS:
Overall Officials: Colleen Kraft, MD, MSc, Principal Investigator — Emory University
Locations (3):
- United States (3):
  - Emory Clinic, Atlanta, Georgia
  - Emory Hospital, Atlanta, Georgia
  - The Hope Clinic of the Emory Vaccine Center, Decatur, Georgia